CLINICAL TRIAL: NCT01905189
Title: Resynchronisation Therapy of Right Ventricle in Pulmonary Arterial Hypertension
Acronym: RETRIEVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A01612-41
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; cardiac resynchronization therapy
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hemodynamic study, cardiac pacing (Experimental): We propose to study the hemodynamic response to a temporary atrio-dual right ventricular stimulation in pulmonary arterial hypertension subjects.Patients will be is own comparator.
  Interventions: Procedure: Resynchronization therapy of right ventricle

INTERVENTIONS:
Procedure: Resynchronization therapy of right ventricle — Right atrio-ventricular resynchronization therapy combined with right intra-ventricular resynchronization therapy

SUMMARY:
Pulmonary arterial hypertension is a disease characterised by pathological changes in the pulmonary arteries leading to a progressive increase in pulmonary vascular resistance and pulmonary artery pressure. Right ventricular failure is the main cause of death in patients with pulmonary arterial hypertension, and the ability of the right ventricle to adapt to the progressive increase in pulmonary vascular resistance associated with changes to the pulmonary vasculature in pulmonary arterial hypertension is the main determinant of a patient's functional capacity and survival.

Right ventricular dyssynchrony was present in a substantial proportion of patients with pulmonary arterial hypertension and this dyssynchrony adversely affected right ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension type I, III, IV, V Dana Point classification
* NYHA classification equal or superior to stage II
* During right catetherization : cardiac index inferior or equal 2.5 L/mn/m2 and atrial pressure superior or equal 10 mmHg OR cardiac index equal or inferior to 2.2 L/mn/m2
* Optimal therapy considered by the referring specialist practioner of the patient

Exclusion Criteria:

* Minor or incapacitated adult
* Pregnancy
* Unability to give free and informed consent
* Pulmonary hypertension type II Dana Point classification
* Eisenmenger syndrome
* Patent foramen ovale
* Left bundle-brach block
* Pulmonary hypertension exacerbation
* Medical clinical situation considered inappropriate by the investigator
* Patient eligible for a heart-lung transplant
* Patient eligible for pulmonary endarterectomy
* Patient with poor echogenicity
* Filter in the inferior vena cava

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
cardiac index measured during right catheterization | After two minutes of right stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Ursmar Milliez, Principal Investigator — Caen UH
Locations (1):
- Caen UH, Caen, Basse-Normandie, France